CLINICAL TRIAL: NCT00143585
Title: Multicentre, Randomized,Double Blind,Placebo Controlled Trial of Myocardial Angiogenesis Using VEGF165, Intramyocardial Gene Delivery in Patients With Severe Angina
Brief Title: NOGA Angiogenesis Revascularization Therapy: Evaluation by RadioNuclide Imaging - The Northern Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-065
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Myocardial Ischemia
Keywords: angiogenesis; VEGF
MeSH Terms: conditions — Myocardial Ischemia

INTERVENTIONS:
Procedure: intramyocardial delivery of either VEGF165 or placebo

SUMMARY:
To demonstrate the clinical efficacy and safety of vascular endothelial growth factor(VEGF165)when delivered by direct myocardial injection through the NOGA navigational catheter to improve myocardial perfusion in patients with severe angina pectoris for whom conventional PCI or CABG are either not possible or not ideal.Secondary objective will be to determine the effects of VEGF gene therapy on angina symptoms, patient perceived quality of life and exercise capacity

DETAILED DESCRIPTION:
A multicentre, double blind, placebo controlled trial to assess efficacy of VEGF and promote myocardial angiogenesis in patients with CCS III-IV angina symptoms,treated with maximal anti anginal medications who are not amenable to or not ideal candidates for conventional revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Canadian Cardiovascular Class III-IV angina despite treatment with maximal medical therapy
* LVEF>20%
* Ischemic defects on myocardial stress SPECT imaging

Exclusion Criteria:

* NYHA>2
* History of or diagnosis of age related macular degeneration, retinopathy
* Atrial fibrillation
* Primary valvular heart disease
* Evidence of or known history of cancer with in past 10 yea
* Uncontrolled hypertension
* Liability to receive dipyridamole
* History or diagnosis of rheumatoid arthritis
* Recent MI(within 4 weeks)
* Important ilio-femoral peripheral vascular disease, limiting catheter access
* History of unexplained gastrointestinal hemorrhage with the past 5 years
* LV thrombus visualized by either echocardiography or contrast LV angiogram
* Other severe concurrent illnesses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-06; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Myocardial perfusion-stress/ rest scores(SRS),changes in summed stress scores(SSS)from baseline to 12 weeks follow up between placebo and VEGF treated groups. This analysis will be repeated at 6 months

SECONDARY OUTCOMES:
symptom evaluation (CCS class, Seattle Angina Questionnaire; patient perceived Quality of Life( SF 36 questionnaire); exercise performance; major adverse cardiac events

CONTACTS AND LOCATIONS:
Overall Officials: Duncan J. Stewart, MD, Principal Investigator — Unity Health Toronto
Locations (7):
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institute de Cardiologie, Hopital Laval, Québec, Quebec